CLINICAL TRIAL: NCT05976347
Title: Identifying and Treating Depression in the Orthopaedic Trauma Population
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00096491; MSKRSH040123 (Other: Atrium Health)
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Fluoxetine; Duloxetine Hydrochloride; Observation; Health Resources

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive either an Selective serotonin reuptake inhibitors (SSRI) or serotonin and norepinephrine reuptake inhibitors (SNRI), and patients who are not interested in taking medication for their symptoms will be enrolled in an observational arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Selective serotonin reuptake inhibitors (SSRI) (Experimental): Fluoxetine, 20mg once daily
  Interventions: Drug: Fluoxetine 20 MG
- serotonin and norepinephrine reuptake inhibitors (SNRI) (Experimental): Duloxetine, 30mg once daily
  Interventions: Drug: Duloxetine 30 MG
- Observational (Other): Referral to behavioral health per standard practice and provision of resources for strategices to address depressive symptoms.
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Fluoxetine 20 MG — Fluoxetine 20 mg once daily
  Other Names: Prozac Weekly, Sarafem, Prozac
  Arms: Selective serotonin reuptake inhibitors (SSRI)
Drug: Duloxetine 30 MG — Duloxetine 30 mg once daily
  Other Names: Irenka and Cymbalta
  Arms: serotonin and norepinephrine reuptake inhibitors (SNRI)
Other: Observation — Referral to behavioral health and resources for addressing depressive symptoms
  Other Names: Referral to behavioral health and resources
  Arms: Observational

SUMMARY:
The goal of this trial is to pilot a way for orthopaedic surgeons to safely screen for depression and provide treatment for depression with medication. The main questions it aims to answer are:

1. What are the outcomes of patients who screen positive for depressive symptoms and are prescribed either an Selective serotonin reuptake inhibitors (SSRI) or serotonin and norepinephrine reuptake inhibitors (SNRI).
2. What are the outcomes of patients who screen positive for depressive symptoms and choose not to pursue treatment with medication?

DETAILED DESCRIPTION:
Depression is common among orthopaedic trauma patients and associated with worsened outcomes including pain, opioid consumption, patient-reported outcomes ,complications, and length of stay. Addressing depression, therefore, should lead to improved outcomes. Orthopaedic surgeons may believe treating depression is outside their scope or that they lack tools to address depressive symptoms. In fact, only 45% of surgeons report they are likely to screen patients, and only 27% are likely to refer patients for psychological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to an Orthopaedic trauma clinic for the first time following operative extremity fracture or any pelvis fracture
* A score of greater than or equal to 5 on the Patient Health Questionnaire-9 (PHQ-9) at first post- operative visit
* Age 18 or older
* Speak English or Spanish

Exclusion Criteria:

* Currently taking medication to treat depression
* Contraindication/allergy to one of the study medications
* Bipolar disorder of psychotic disorder
* Endorse suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptom Scores | Baseline
  Improvement in depressive symptoms, indication by either remission (PHQ-9 score <5) or a 50% reduction in PHQ-9 score. The Patient Health Questionnaire (PHQ-9) is a self-report tool that incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms. The too rates the frequency of the symptoms which factors into the scoring severity index. PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe and severe depression.
Depressive Symptom Scores | Month 3
  Improvement in depressive symptoms, indication by either remission (PHQ-9 score <5) or a 50% reduction in PHQ-9 score. The Patient Health Questionnaire (PHQ-9) is a self-report tool that incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms. The too rates the frequency of the symptoms which factors into the scoring severity index. PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe and severe depression.
Depressive Symptom Scores | Month 6
  Improvement in depressive symptoms, indication by either remission (PHQ-9 score <5) or a 50% reduction in PHQ-9 score. The Patient Health Questionnaire (PHQ-9) is a self-report tool that incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms. The too rates the frequency of the symptoms which factors into the scoring severity index. PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe and severe depression.
Depressive Symptom Scores | Month 9
  Improvement in depressive symptoms, indication by either remission (PHQ-9 score <5) or a 50% reduction in PHQ-9 score. The Patient Health Questionnaire (PHQ-9) is a self-report tool that incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms. The too rates the frequency of the symptoms which factors into the scoring severity index. PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe and severe depression.
Depressive Symptom Scores | Year 1
  Improvement in depressive symptoms, indication by either remission (PHQ-9 score <5) or a 50% reduction in PHQ-9 score. The Patient Health Questionnaire (PHQ-9) is a self-report tool that incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms. The too rates the frequency of the symptoms which factors into the scoring severity index. PHQ-9 scores of 5, 10, 15, and 20 represent mild, moderate, moderately severe and severe depression.

SECONDARY OUTCOMES:
Adherence to Treatment Percentage | Months 3, 6, and 12
  Adherence to treatment and side effects or adverse events associated with the medications will be collected using patient logs, study visit questionnaires, and the medical record (i.e., number of prescriptions filled).
Utilization of non-pharmaceutical tools and resources Percentage | Months 3, 6, and 12
  Engagement with behavioral health resources will be collected using patient logs, study visit questionnaires, and the medical record (i.e., number of visits with Behavioral Health).
Patient Reported Outcome Measures - PROMIS-29 Scores | Months 3, 6, and 12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores mean a higher level of disability.
Patient Reported Outcome Measures - Work Productivity and Activity Impairment Questionnaire Scores | Months 3, 6, and 12
  The Work Productivity and Activity Impairment questionnaire measures how work productivity and activities are impaired by a specific health condition or disease. Scores are expressed as a percentage of impairment/productivity loss, a high score indicates greater impairment.
Patient Reported Outcome Measures - Brief Pain Inventory Scores | Months 3, 6, and 12
  Assesses the severity of pain and the impact of pain on daily functions. Assesses the severity of and impact of pain on daily function. Patients are asked to rate their current symptoms, average experiences of pain, and the minimum and maximum intensities of their symptoms on scales that range from 1-10. A total pain severity score can be found by averaging these items or a single items can be treated as the primary outcome. Higher scores indicate greater severity and more interference.
Healthcare Utilization - The number of hospitalizations and ED visits | Months 3, 6, and 12
  The number of hospitalizations and ED visits
Patient Reported Outcome Measures: Patient Health Questionnaire 9 (PHQ-9) | Months 3, 6, and 12
  A PHQ-9 score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression. The higher the score, the more symptoms of depression experienced, and the more severe the depression is.
Patient Reported Outcome Measures - Veterans RAND 12 Item Health Survey (VR-12) | Months 3, 6, and 12
  Measures health related quality of life across 7 domains. The answers are summarized into two scores - a Physical Component Score and a Mental Component Score.
Qualitative Interview Information | One time between 6-12 months
  Patients in the observational arm will participate in semi-structured interviews. Interviews will be recorded and transcribed verbatim within one week. Field notes will be written within one week of each interview, and the interview guide will be revised as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan K Wally, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No